CLINICAL TRIAL: NCT06540456
Title: Qutenza 8% Capsaicin Topical System for the Treatment of Neuropathic Axial Lower Back Pain and Lumbosacral Radiculopathy: a Prospective Study.
Brief Title: Qutenza 8% Capsaicin Topical System for the Treatment of Neuropathic Axial Lower Back Pain and Lumbosacral Radiculopathy
Status: Enrolling by invitation | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Collaborators: Averitas Pharma, Inc. (Industry)
Responsible Party: Principal Investigator, Matthew Sherrier, Assistant Professor-Faculty, Medical University of South Carolina
Other Study IDs: Pro00134392
Record Dates: First submitted 2024-06-28; First posted 2024-08-06 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Lower Back Pain; Lumbosacral Radiculopathy
MeSH Terms: conditions — Low Back Pain | interventions — Capsaicin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Patients with neuropathic LBP and painful lumbosacral radiculopathy: patients with neuropathic LBP and painful lumbosacral radiculopathy
  Interventions: Drug: Qutenza® 8% Capsaicin Topical System

INTERVENTIONS:
Drug: Qutenza® 8% Capsaicin Topical System — Treatment of patients with neuropathic LBP and painful lumbosacral radiculopathy using the Qutenza 8% capsaicin topical system.

SUMMARY:
This is a research study to find out if Qutenza 8% capsaicin topical system is safe and effective when treating subjects with lower back pain (LBP) that is caused by damage at or near the nerve's root in the lower back leg (lumbosacral radiculopathy) which is pain that can move all the way down the back of the leg. The pain may also start outside of the spinal cord, in the peripheral nerves and may also be felt all the way down the back of the leg (neuropathic LBP). Qutenza 8% capsaicin, the study drug, is currently FDA approved to treat nerve pain after a shingles outbreak in addition to a type of nerve pain in the feet associated with diabetes. In this study a maximum of four patches per visit (sized 14cm x 20 cm) will be used to deliver the Qutenza 8% capsaicin to the participants skin.

If a subject meets the qualifications for this study, in addition to their standard of care for their LBP, they can expect to have a total of 5 visits in a 12 month period. Each visit will require subjects to fill out several surveys and receive treatment patches for their LBP (your doctor will decide if participants will need to be retreated at each visit based on your symptoms). The study visits are estimated to take 90 minutes upwards to 120 minutes.

DETAILED DESCRIPTION:
Chronic lower back pain (LBP) and lumbosacral radiculopathy are common, disabling, and costly conditions. The lifetime prevalence of LBP is estimated to be greater than 70% in industrialized countries, with a 1-year prevalence of 15-45% and LBP is the most common cause of years lived with disability worldwide. Chronic LBP (defined as LBP lasting less than 3 months) is a complex and heterogeneous condition with nociceptive and neuropathic components.

The goals of treatment of chronic LBP and lumbosacral radiculopathy are to reduce pain, maintain function, and prevent future exacerbation. Guidelines advocate for a multimodal approach to the management of these conditions, combining pharmacological therapies for symptomatic relief with nonpharmacological approaches, such as physical rehabilitation. Choice of treatment is individualized according to the nature and severity of symptoms, the presence of comorbid conditions, potential for adverse effects and drug interactions, and cost. At this time, there are no specific recommendations for treatment of the neuropathic components of chronic LBP and neuropathic pain medications for painful radiculopathy have limited response rates. Furthermore, current pharmacologic approaches for the treatment of neuropathic pain are associated with a risk of significant adverse effects, which can have a serious impact on patients' quality of life. As such, there is a pressing need for safe and effective therapeutic options in treating neuropathic LBP and painful lumbosacral radiculopathy.

Capsaicin is the main compound in chili peppers and acts mechanistically as a selective agonist of the transient receptor potential vanilloid 1 (TRPV1) channel, which is highly expressed on nociceptors. High concentrations of capsaicin have been effectively utilized for the treatment of neuropathic pain. Additionally, whereas many pharmacologic and interventional pain relief options for chronic LBP and radiculopathy cause weight gain, capsaicin has been widely studied for its weight loss potential.

Emerging evidence suggests the use of topical capsaicin may be a safe and efficacious treatment for chronic LBP and radiculopathy. With regards to LBP, a 2010 double-blind multi-center randomized clinical trial on the use of 0.05% topical capsaicin cream for the treatment of chronic LBP demonstrated a significantly higher number of patients experiencing at least 50% pain sum score improvement at 3 weeks compared to placebo. A 2016 open-label study of 90 patients with lumbosacral neuropathic pain who received treatment with a topical 8% capsaicin patch found statistically significant reductions in pain at 2, 8, and 12 weeks follow-up. With regards to lumbosacral radiculopathy, a 2017 randomized controlled trial of 50 participants with chronic lumbosacral radiculopathy treated with a topical 8% capsaicin patch found at least a 30% improvement of pain in 71.4% and 39.1% of patients with 3 months to 2 years duration of pain and greater than 2 years duration of pain, respectively. A prospective study investigating the use of a single 8% capsaicin patch in patients with a variety of neuropathic pain conditions, including radiculopathy noted that the proportions of patients achieving a 30% and 50% decrease in pain at 12 weeks were 43% and 24%, respectively. Additionally, a small retrospective analysis of patients with painful radiculopathy found that the capsaicin 8% patch provided rapid and sustained pain relief, with a significant reduction in prescribed concomitant pain medications. In brief, the current literature is limited by small sample sizes and short follow up periods but does suggest topical capsaicin is a rational choice for the treatment of neuropathic lumbosacral pain.

The neuropathic components in chronic LBP and lumbosacral radiculopathy may be under-recognized and therefore undertreated. Most clinical trials of drug treatments for neuropathic pain have examined patients with Postherpetic neuralgia or painful diabetic peripheral neuropathy, and the extent to which results of these studies can be extrapolated to other neuropathic conditions is unknown. Use of the Qutenza (8% capsaicin) topical patch for the treatment of chronic LBP and lumbosacral radiculopathy holds great promise to improve the pain and function of patients suffering with these common and debilitating conditions, which in turn has the potential for tremendous economic impact.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years of age
* Willing and have capacity to provide informed consent
* History of symptoms for longer than three months (so as to minimize the chance of spontaneous recovery)
* Pain-DETECT questionnaire (PD-Q) indicating neuropathic component of pain

Exclusion Criteria:

* Self-reported or medical records showing history of lumbar spine, hip, or lower extremity surgeries within three months
* Chronic opioid use (determined by self-report and review of Prescription Drug Monitoring Program database) - defined as more than 15 morphine milligram equivalents (MME) per day for at least 2 weeks
* Self-reported or medical records showing history of painful peripheral neuropathies (from diabetes mellitus, HIV, or induced by chemotherapy)
* Self-reported allergies to study medications
* Pregnant women (determined by self-report) and prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the Physical Medicine and Rehabilitation clinics at the Medical University of South Carolina outpatient clinics with complaints of lower back pain and radicular leg pain who meet all inclusion and exclusion criteria will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2027-07-03 (Estimated); Study Completion 2028-07-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse effects as assessed by routine patient monitoring of subjects treated with Qutenza 8% capsaicin topical system for LBP and lumbosacral radiculopathy | at 12 months
  The primary aim of this pilot study is to assess whether the Qutenza 8% capsaicin topical system is an effective treatment for neuropathic lower back pain and painful lumbosacral radiculopathy as based on PROMIS-29 scores for pain and quality of life. Safety will be determined by the number of participants with treatment-related adverse events as assessed by routine clinical monitoring

SECONDARY OUTCOMES:
Assess changes in body mass index (BMI) in patients receiving the Qutenza 8% capsaicin topical system. | at 12 months
  A secondary aim is to assess side effects, weight (measured in kg) and height (measured in meters) will be combined to report changes in BMI in kg/m^2 at each subsequent follow-up visit of patients receiving the Qutenza 8% capsaicin topical system.
Assess changes in quality of life and sleep in patients receiving the Qutenza 8% capsaicin topical system. | at 12 months
  A secondary aim is to assess the quality of life and sleep data will be obtained from the PROMIS 29 subscales
Assess changes in medication and procedural utilization in patients receiving the Qutenza 8% capsaicin topical system. | at 12 months
  A secondary aim is to assess medication and procedural (lumbar and sacral interventions, including sacroiliac joint injections or radiofrequency ablations, lumbar facet joint injections or radiofrequency ablation, and lumbar or sacral epidural steroid injections) utilization, which will be determined by patient's self-report interview or chart review at each subsequent follow-up visit of patients receiving the Qutenza 8% capsaicin topical system.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Sherrier, Principal Investigator — Medical University of South Carolina
Locations (1):
- MUSC Health Nexton Medical Park, Summerville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No